CLINICAL TRIAL: NCT00584168
Title: Decreasing Morbidity After Uvulopalatopharyngoplasty With the Use of Dexamethasone - A Randomized Double Blinded Placebo Controlled Trial
Brief Title: Using Dexamethasone After Uvulopalatopharyngoplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dexamethasone, UPPP - Houck; UPPP Study, IRB # 12098 (Other: Institutional Review Board)
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Pain
Keywords: UPPP; Dexamethasone; Uvulopalatopharyngoplasty; Pain Management; Increasing pain management in patients that have undergone UPPP surgery
MeSH Terms: conditions — Pain; Agnosia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Patient will receive a placebo.
  Interventions: Drug: Placebo
- 1 (Experimental): Patient will receive dexamethasone.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — They will take a pill the day before surgery, twice daily for the next four days and then once daily for the next two days for a total of seven days.
  Arms: 1
Drug: Placebo — They will take a pill the day before surgery, twice daily for the next four days and then once daily for the next two days for a total of seven days.
  Arms: 2

SUMMARY:
This study looks at lessening the pain after a Uvulopalatopharyngoplasty (UPPP) surgery by using Dexamethasone (a corticosteroid).

DETAILED DESCRIPTION:
The study was designed because patients have a lot of pain after they have a UPPP. Certain drugs called steroids may lessen the pain associated from this surgery. This study uses Dexamethasone (a corticosteroid), to see if it will help reduce pain, decrease the amount of time until the patient can begin to eat or return to normal activity, or increase their satisfaction with pain management. In this study the patients will be randomized (computer chosen) to receive either the study drug (dexamethasone), or a placebo. The patient will start the day before surgery with a single pill. They will then receive the dexamethasone or a placebo twice daily for the next four days and then once daily for the next two days for a total of seven days. Afterward, they will be asked to complete a questionnaire. The five questions ask patients to access the amount of pain they have, how much of their normal diet or activity they have returned to, and how much pain medication they have taken. At the next follow-up visit they will be asked to complete another questionaire (9 questions) about the patient's satisfaction with pain management.

ELIGIBILITY:
Inclusion Criteria:

* Candidates scheduled for UPPP surgery.
* Able to take steroids

Exclusion Criteria:

* Those patients who unable to take steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Quantifying patient treatment with a questionaire. Patient will rate their satisfaction with pain management. | Eleven days post-operative

CONTACTS AND LOCATIONS:
Overall Officials: John Houck, MD, Principal Investigator — University of Oklahoma
Locations (2):
- United States (2):
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center, Oklahoma City, Oklahoma